CLINICAL TRIAL: NCT07059936
Title: Predicting Immunotherapy Response and Survival of Liver Cancer Patients Using Artificial Intelligence and Radiomics (Radiology-AI-Liver)
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0620
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CT imaging data and MR imaging data from liver cancer (hepatocellular carcinoma) patients prior to the initiation of immunotherapy (and possibly also after treatment) will be collected. The processing pipeline includes automatic tumor segmentation, radiomics feature extraction, feature selection, and construction of a classification model.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were treated for hepatocellular carcinoma in Wuhan Union Hospital from July 2025 to July 2026;
2. Aged > 18 years old;
3. At least one CT scan or MR scan before treatment;
4. Tissue biopsy pathological examination confirmed the diagnosis of the above tumors.

Exclusion criteria:

1. Poor image quality;
2. Incomplete clinical data or loss of follow-up;
3. Presence of another primary malignancy other than liver cancer;
4. Unclear pathological diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 1 year
Progression-free survival | 1 year
overall survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei, China